CLINICAL TRIAL: NCT03338101
Title: Comparative Study Between the Goldmann Flattening Tonometer and the Non-Contact Tonometer in Patients of a Reference Ophthalmological Hospital
Brief Title: Comparative Study Between Tonometers
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: TRABALHO GLENDA ARVO 2018
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Glaucoma Eye

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comparative study between the Goldmann Flattening Tonometer and the Non-Contact Tonometer in patients of a Reference Ophthalmological Hospital

ELIGIBILITY:
Inclusion Criteria:Pacients with glaucoma diagnosed -

Exclusion Criteria:Pacients without glaucoma diagnosed

-

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with glaucoma diagnosed who are monitorated in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Comparative study between the Goldmann Flattening Tonometer and the Non-Contact Tonometer in patients of a Reference Ophthalmological Hospital | 3 months
  evaluation of the intraocular pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No